CLINICAL TRIAL: NCT05188638
Title: Single-centre, Randomised, Placebo-controlled, and Double-blinded First-in-human Clinical Study Investigating the Safety and Tolerability of Ascending Single and Multiple Doses of Nebulised SoftOx Inhalation Solution in Healthy Subjects
Brief Title: Safety of Ascending Single and Multiple Doses of Nebulised SoftOx Inhalation Solution in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: SoftOx Solutions AS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SIS-01; 2020-004462-19 (EudraCT Number)
Record Dates: First submitted 2021-12-09; First posted 2022-01-12 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Healthy Volunteers; Safety

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Single dose of up to 5 mL nebulised SIS @ 25 ppm/placebo (Experimental)
  Interventions: Drug: SoftOx Inhaled Solution (SIS); Drug: Placebo
- Single dose of up to 5 mL nebulised SIS @ 50 ppm/placebo (Experimental)
  Interventions: Drug: SoftOx Inhaled Solution (SIS); Drug: Placebo
- Single dose of up to 5 mL nebulised SIS @ 100 ppm/placebo (Experimental)
  Interventions: Drug: SoftOx Inhaled Solution (SIS); Drug: Placebo
- OD dosing of up to 5 mL nebulised SIS @ x ppm/placebo for 5 days (Experimental): The dose to be administered in the multiple dose groups will depend on the results obtained in the single dose groups and will be decided by the SMC. The dose tested in the first multiple dose group will be the second highest well-tolerated single dose or lower.
  Interventions: Drug: SoftOx Inhaled Solution (SIS); Drug: Placebo
- OD dosing of up to 5 mL nebulised SIS @ y ppm/placebo for 5 days (Experimental)
  Interventions: Drug: SoftOx Inhaled Solution (SIS); Drug: Placebo
- BID dosing of up to 5 mL nebulised SIS @ y ppm/placebo, for 4 days + morning dose on Day 5 (Experimental)
  Interventions: Drug: SoftOx Inhaled Solution (SIS); Drug: Placebo
- QID dosing of up to 5 mL nebulised SIS @ y ppm/placebo for 4 days + morning dose on Day 5 (Experimental)
  Interventions: Drug: SoftOx Inhaled Solution (SIS); Drug: Placebo

INTERVENTIONS:
Drug: SoftOx Inhaled Solution (SIS) — SIS consists of the active compound, hypochlorous acid (HOCl). Concentrations of SIS refer to the concentration of HOCl in parts per million (ppm).
Drug: Placebo — Sterile isotonic saline

SUMMARY:
Background:

This first-in-human study will investigate the safety and tolerability of single and multiple doses of nebulised SoftOx Inhalation Solution (SIS) delivered via a jet nebuliser to healthy subjects.

Objectives:

The objective of the current study is to assess the safety and tolerability of single and multiple ascending doses of nebulised SIS in healthy subjects.

Eligibility:

Subjects are eligible to participate in this study if they are healthy, between 18 and 55 years of age, and have a Body Mass Index (BMI) of ≥ 18.5 and ≤ 29.9 kg/m2.

Subjects are not eligible to participate in this study if they have recently participated in another clinical trial or have donated blood, have a medical condition or a history of drug hypersensitivity, are using concomitant medication, or have a positive drugs of abuse test.

Design:

A randomised, double-blind, and placebo-controlled trial. Subjects will be enrolled into one of three single dose groups or into one of four multiple dose groups. The two first multiple dose groups will be dosed once daily (OD) for five days. The two last multiple dose groups will be dosed twice daily (BID) for four days plus a morning dose on Day 5, or four times daily (QID) for four days plus a morning dose on Day 5, respectively.

The investigational medicinal product (SIS or placebo; IMP) will be delivered via a jet nebuliser and inhaled through a mask over a period of up to 15 minutes.

Each treatment group will comprise eight subjects who will be randomised to receive SIS or placebo in a 3:1 ratio.

A Safety Monitoring Committee (SMC) will review the safety and tolerability data from all preceding groups and decide whether the planned next dose regimen is acceptable prior to initiating the dosing in a new dose group.

The dose to be administered in the multiple dose groups will depend on the results obtained in the single dose groups and will be decided by the SMC. The dose tested in the first multiple dose group will be the second highest well-tolerated single dose or lower.

ELIGIBILITY:
Inclusion Criteria:

1. Has signed a written informed consent.
2. Is 18 to 55 years of age (both inclusive). Women of child-bearing potential must be sexually abstinent or should agree to use effective contraceptive methods3 throughout the course of the study.
3. Has a Body Mass Index (BMI) of 18.5-29.9 kg/m2 (both inclusive).
4. Good health in the opinion of the Investigator based upon medical history, physical examination, vital signs, oxygen saturation, electrocardiogram (ECG), lung function, and laboratory profile of blood and urine.
5. Is able to comply with the inhalation procedure of inhaling through the nose and exhaling through the mouth, in the opinion of the Investigator.
6. Has negative urine drug screen and negative alcohol breath test on the day of screening and before the (first) administration of IMP.

Exclusion Criteria:

1. Any surgical or medical condition, including findings in the medical history or in the pre-study assessments, or any other significant disease, that in the opinion of the Investigator, constitutes a risk or a contraindication for the participation of the subject in the study or that could interfere with the study objectives, conduct, or evaluation.
2. Has had cancer within the last 10 years except for adequately managed basal cell carcinoma and squamous cell carcinoma of the skin.
3. Intake of any prescription or non-prescription medication, or herbal products with known pharmacological effects (e.g., St. John's wort), within 2 weeks or 5 half-lives of the drug, whichever is longer, before the (first) administration of IMP with the exception of paracetamol, which is allowed up to 1000 mg QID dosed according to labelling as well as hormonal contraceptives and hormonal replacement therapy.
4. Participation in the treatment phase of a clinical trial with an investigational new drug within one month before the (first) administration of IMP.
5. Is a smoker or has used any form of nicotine product including e-cigarette, snuff, chewing tobacco, nicotine gum, etc., on a regular basis within three months before the (first) administration of IMP.
6. Has a history (within the last two years) or is at present an abuser of alcohol or narcotics, or is a user of recreational drugs (e.g., cocaine).
7. Has donated or lost > 400 mL blood within one month before the (first) administration of IMP.
8. Has previously been randomised in this study.
9. Is pregnant or lactating at screening or time of the (first) administration of IMP.
10. Ascertained or presumptive allergy/hypersensitivity to SIS; history of anaphylaxis to drugs or serious allergic reactions leading to hospitalization or any other allergy reaction in general, which the Investigator considers may affect the safety of the subject and/or outcome of the study.
11. Inability to communicate or cooperate with the Investigator (e.g., language problem, illiteracy, poor mental status) or to comply with the requirements of the study.
12. Legal incapacity or limited legal capacity.
13. Is considered by the Investigator, unsuitable to participate in the study for any other reason.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2022-04-13 (Actual); Study Completion 2022-04-13 (Actual)

PRIMARY OUTCOMES:
Occurrence of adverse events (AEs). | From the start of the first administration of IMP to 2 or 3 days after the last administration of IMP
Severity of adverse events (AEs). | From the start of the first administration of IMP to 2 or 3 days after the last administration of IMP
Change from baseline in forced expiratory volume in 1 second (FEV1) | From 30 minutes after the start of the first administration of IMP to 2 or 3 days after the last administration of IMP
Change from baseline in oxygen saturation measured by pulse oximetry | From the start of the first administration of IMP to 2 or 3 days after the last administration of IMP
Change from baseline in local tolerability | Immediately after completion of the inhalation to 2 or 3 days after the last administration of IMP
  Subjects will be asked to complete a brief questionnaire regarding symptoms (irritation, burning sensation/pain, coughing, sneezing, or other) from the mouth, nose, and respiratory tract.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M Burton, MD; PhD, Study Director — SoftOx Solutions A/S; David P Sonne, MD; PhD, Principal Investigator — Bispebjerg Hospital
Locations (1):
- DanTrials ApS, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No